CLINICAL TRIAL: NCT00003556
Title: Phase Ib Trial of Intratumoral Injection of a Recombinant Canarypox Virus Encoding Human B7.1 (ALVAC-hB7.1) or a Combination of ALVAC-hB7.1 and a Recombinant Canarypox Virus Encoding Human Interleukin 12 (ALVAC-hIL-12) in Patients With Surgically Incurable Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02274; UAB-9705; NCI-T97-0046; CDR0000066619 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-08-17 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Arm I (Experimental): Patients receive ALVAC-hB7.1 alone or combined with ALVAC-hIL-12 intratumorally on days 1, 4, 8, and 11. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated at each dose level of ALVAC-hB7.1. The maximum tolerated dose is defined as the dose of ALVAC-hB7.1 at which no more than 1 of 5 patients experiences dose limiting toxicity.
  Interventions: Biological: ALVAC-hB7.1; Biological: canarypox-hIL-12 melanoma vaccine

INTERVENTIONS:
Biological: ALVAC-hB7.1
Biological: canarypox-hIL-12 melanoma vaccine

SUMMARY:
Phase I trial to study the effectiveness of vaccine therapy in treating patients with melanoma that cannot be treated with surgery. Vaccines may make the body build an immune response that may kill tumor cells. Combining more than one vaccine may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxic effects associated with ALVAC-hB7.1 alone or combined with ALVAC-hIL-12 in patients with surgically incurable melanoma.

II. Characterize the inflammatory and lymphokine response to this regimen in these patients.

III. Examine the extent of nodule regression, humoral immune response, and cytolytic T cell activity with this regimen in these patients.

OUTLINE: This is a dose escalation study of ALVAC-hB7.1

Patients receive ALVAC-hB7.1 alone or combined with ALVAC-hIL-12 intratumorally on days 1, 4, 8, and 11. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated at each dose level of ALVAC-hB7.1. The maximum tolerated dose is defined as the dose of ALVAC-hB7.1 at which no more than 1 of 5 patients experiences dose limiting toxicity.

Patients are followed at 1, 2, 4, 8, 11, 15, 22, and 43 days after the first vaccination.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma that is surgically incurable
* At least one dermal, subcutaneous or lymph node metastasis that is evaluable for local response and accessible for injection
* If only one accessible lesion is available, it must be at least 2 cm
* If two or more accessible lesions exist, then none of them are required to be at least 2 cm

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-2
* Life expectancy: Greater than 3 months
* Leukocyte count at least 3,000/mm3
* Platelet count at least 120,000/mm3
* SGOT and alkaline phosphatase less than 5 times normal
* Bilirubin less than 1.5 mg/dL (unless secondary to hepatic metastasis)
* BUN less than 40 mg/dL
* Creatinine less than 2.5 mg/dL
* No evidence of congestive heart failure, unstable angina, or serious cardiac arrhythmias
* Not positive for hepatitis B virus
* Not positive for HIV
* No history of allergy to vaccinia virus
* No evidence of other primary tumors except for basal cell carcinoma, squamous cell skin carcinoma, or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No underlying immunodeficiency disorder

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior biologic therapy (e.g., interferon or IL-2)
* At least 30 days since prior chemotherapy
* No concurrent steroids
* At least 30 days since prior radiotherapy
* Prior radiotherapy to no greater than 50% of nodal groups
* No prior splenectomy
* No concurrent drugs which affect immune function (e.g., glucocorticoids or cimetidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1999-01; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Conry, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States